CLINICAL TRIAL: NCT03244020
Title: Low Molecular Weight Heparin Versus Aspirin for Venous Thromboembolism Prophylaxis in Orthopaedic Oncology
Brief Title: LMWH vs Aspirin for VTE Prophylaxis in Orthopaedic Oncology
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Johns Hopkins University (Other); University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Santiago Lozano-Calderon, Associate Professor of Orthopaedic Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017P000382
Record Dates: First submitted 2017-08-05; First posted 2017-08-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Sarcoma; Soft Tissue Sarcoma; Bone Sarcoma; Bone Metastases; Venous Thromboembolism; Hematoma; Anticoagulant-induced Bleeding
MeSH Terms: conditions — Sarcoma; Bone Neoplasms; Venous Thromboembolism; Hematoma | interventions — Aspirin; Enoxaparin

STUDY DESIGN:
Intervention Model Description: Three separate patient categories are being investigated in this trial. All patients are undergoing pelvic and/or lower extremity surgery for one of three possible conditions: 1) soft tissue sarcoma; 2) primary bone sarcoma; 3) metastatic bone disease. Within each of these groups, patients will be randomized to either aspirin or low molecular weight heparin (enoxaparin) for venous thromboembolism prophylaxis post operatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- LMWH for Soft Tissue Sarcoma (Experimental): Patients undergoing surgery for pelvic/lower extremity soft tissue sarcomas and are randomized to Enoxaparin 40Mg/0.4mL prefilled syringe subcutaneous injection daily for VTE prophylaxis
  Interventions: Drug: Enoxaparin 40Mg/0.4mL Prefilled Syringe
- ASA for Soft Tissue Sarcoma (Experimental): Patients undergoing surgery for pelvic/lower extremity soft tissue sarcomas and are randomized to aspirin 325 mg po daily for VTE prophylaxis
  Interventions: Drug: Aspirin 325mg
- LMWH for Primary Bone Tumor (Experimental): Patients undergoing surgery for pelvic/lower extremity primary bone tumor and are randomized to Enoxaparin 40Mg/0.4mL prefilled syringe subcutaneous injection daily for VTE prophylaxis
  Interventions: Drug: Enoxaparin 40Mg/0.4mL Prefilled Syringe
- ASA for Primary Bone Tumor (Experimental): Patients undergoing surgery for pelvic/lower extremity primary bone tumor and are randomized to aspirin 325 mg po daily for VTE prophylaxis
  Interventions: Drug: Aspirin 325mg
- LMWH for Metastatic Disease (Experimental): Patients undergoing surgery for pelvic/lower extremity metastatic bone disease and are randomized to Enoxaparin 40Mg/0.4mL prefilled syringe subcutaneous injection daily for VTE prophylaxis
  Interventions: Drug: Enoxaparin 40Mg/0.4mL Prefilled Syringe
- ASA for Metastatic Disease (Experimental): Patients undergoing surgery for pelvic/lower extremity metastatic bone disease and are randomized to aspirin 325 mg po daily for VTE prophylaxis
  Interventions: Drug: Aspirin 325mg

INTERVENTIONS:
Drug: Aspirin 325mg — Aspirin 325 mg by mouth once daily
  Other Names: ASA
  Arms: ASA for Metastatic Disease; ASA for Primary Bone Tumor; ASA for Soft Tissue Sarcoma
Drug: Enoxaparin 40Mg/0.4mL Prefilled Syringe — Enoxaparin 40 mg subcutaneous injection once daily
  Other Names: Lovenox
  Arms: LMWH for Metastatic Disease; LMWH for Primary Bone Tumor; LMWH for Soft Tissue Sarcoma

SUMMARY:
Aspirin and low molecular weight heparin (LMWH) are both commonly employed pharmacologic methods of venous thromboembolism (VTE) prophylaxis after orthopaedic surgery. Data comparing these two methods of VTE prophylaxis in patients undergoing pelvic/lower extremity orthopaedic surgery for malignancy are lacking, however, as compared to the data and guidelines present for VTE chemoprophylaxis after joint arthroplasty and hip fracture surgery. In this clinical trial, our specific aim is to compare the post operative incidence of VTE between patients receiving aspirin and LMWH after pelvic/lower extremity orthopaedic oncology procedures.

DETAILED DESCRIPTION:
Lower extremity orthopaedic surgery and malignancy are both known major risk factors for venous thromboembolism (VTE). Guidelines from high quality data exist with regards to VTE prophylaxis in patients undergoing orthopaedic surgery, particularly joint arthroplasty. Far fewer data are available regarding the efficacy of various methods of pharmacologic VTE prophylaxis in patients undergoing surgery for primary or metastatic musculoskeletal malignancies as malignancy itself is known to confer a hypercoagulable state. The existing data, including published data from our institution, are almost exclusively from retrospective studies. Given the limited external validity of existing guidelines and limitations inherent in applying data from retrospective studies, a randomized, prospective study comparing two of the most common methods of pharmacologic VTE prophylaxis would help to guide clinical care of this patient population. In addition, large dead spaces susceptible to hematoma formation are often created from tumor resections in orthopaedic oncology. Our retrospective data suggest that hematoma formation may be an independent predictor of infection. An important risk of chemical VTE prophylaxis is an increased incidence of bleeding into these dead spaces, leading to hematomas. This illustrates the complexity of selecting a method of VTE prophylaxis in patients at both high risk of VTE and hematoma formation and the need for high quality data to guide clinical decision-making in this patient population.

The specific aim of this study is to compare the post operative incidence of symptomatic deep vein thrombosis (DVT) and pulmonary embolus (PE) between patients who receive low molecular weight heparin (LMWH) versus aspirin for prophylaxis after having undergone pelvic or lower extremity orthopaedic oncology surgery (primary bone sarcomas, soft tissue sarcomas, and metastatic osseous disease).

Our secondary aim is to compare the incidence of hematoma formation and wound complications between these methods of pharmacologic prophylaxis in the aforementioned patient population.

Our hypothesis is that there is no significant difference in the incidence rate of symptomatic DVT/PE in patients administered LMWH versus aspirin for prophylaxis; however there may exist a difference in the rate of wound complications between these prophylaxis methods.

ELIGIBILITY:
Patients will first be evaluated for inclusion in a master observational study with the following inclusion criteria:

1. Age ≥18 years
2. Prior or planned surgery on the pelvis or lower extremity
3. Fulfills one of the following:

   a. Cohort A: Metastatic osseous disease, undergoing: i. Endoprosthetic reconstruction ii. Curettage, cement packing, and fixation with nails, plates, and/or screws iii. Intramedullary nail fixation only b. Cohort B: Primary bone sarcoma, undergoing wide resection, amputation, or reconstruction with endoprosthesis, allograft, or allograft-prosthesis composite (APC).

   c. Cohort C: Primary soft tissue sarcoma ≥5 cm in diameter, undergoing wide resection
4. Anticoagulation therapy was received or is planned.

In addition to fulfilling all the inclusion criteria in Part 1 of this study, participants must also not meet any of the below exclusion criteria in order to be eligible for randomization to either aspirin or LMWH.

Exclusion Criteria:

1. Documented prior history of VTE.
2. Preoperative use of therapeutic or prophylactic chemical anticoagulation at the time of surgery.
3. Documented allergy/adverse reaction to either of the two study drugs.
4. Presence of inferior vena cava (IVC) filter.
5. Known, diagnosed hypercoagulable state (other than malignancy).
6. Inability to receive chemical anticoagulation.
7. Preoperative use of full-strength aspirin 325 mg daily; patients already taking aspirin 81 mg daily will not be excluded.
8. Inability for the patient him/herself to give informed consent due to delirium, dementia, or any other reason.
9. Pregnancy
10. Fear of needles that prevents administration of LMWH.
11. Inability to administer medications via needles.
12. For patients with metastatic osseous disease, a Khorana score of ≥3.

Pregnancy testing, via a urine or blood test, is a routine part of pre-operative laboratory testing in patients scheduled to undergo orthopaedic surgeries. Attending surgeons may also choose to exclude any patient from randomization at their discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2868 (Estimated)
Dates: Start 2018-02-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Venous thromboembolism | Up to 3 or 6 months post operatively for bone/soft tissue sarcomas and metastatic osseous disease, respectively
  Deep venous thrombosis; pulmonary embolus

SECONDARY OUTCOMES:
Hematoma formation | Up to 3 or 6 months post operatively for bone/soft tissue sarcomas and metastatic osseous disease, respectively
Complication requiring return to operating room | Up to 3 or 6 months post operatively for bone/soft tissue sarcomas and metastatic osseous disease, respectively
  Return to operating room for any reason related to the original surgery
Early chemoprophylaxis stop | Up to 4 weeks post operatively
  ASA or LMWH stopped prior to 4 weeks post operatively by surgeon for any reason
Infection | Up to 3 or 6 months post operatively for bone/soft tissue sarcomas and metastatic osseous disease, respectively
  Infection requiring any sort of treatment (antibiotics alone, return to operating room)

CONTACTS AND LOCATIONS:
Overall Officials: Santiago A Lozano-Calderon, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (10):
- United States (10):
  - University of California Los Angeles Health, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Louisiana State University Health, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Santiago Lozano-Calderon, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Missouri-Columbia Cancer Care, Columbia, Missouri
  - Cooper University Health Care, Camden, New Jersey
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No